CLINICAL TRIAL: NCT06823284
Title: Characterization of Relative Bioavailability of a Newly Developed Esflurbiprofen Topical System (EFTS) in Comparison with a Marketed Oral Flurbiprofen-containing Tablet Formulation After Multiple-dose Administration Including EFTS Adhesion Assessment - a Phase I, Open-label, Randomized, 2-period, Cross-over Study in Healthy Subjects
Brief Title: To Assess the Bioavailability of TK-254RX in Comparison with Oral Flurbiprofen Tablets and the Adhesion of TK-254RX in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teikoku Seiyaku Co., Ltd. (Industry)
Collaborators: SocraTec R&D GmbH (Other); SocraMetrics GmbH (Industry); HWI pharma services GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TK-254RX-0102; 2024-513058-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-19; First posted 2025-02-12 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — Flurbiprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TK-254RX (Experimental): TK-254RX will be applied to left and right lower leg above ankle once daily over 5 consecutive days i.e. 10 patches will be applied totally.
  Interventions: Drug: Esflurbiprofen Topical System
- Tablet (reference product) (Experimental): Tablets containing 100mg flurbiprofen will be administered three times daily (every 8 h) over 4 consecutive days i.e. 12 tablets will be administered totally.
  Interventions: Drug: Flurbiprofen tablet

INTERVENTIONS:
Drug: Esflurbiprofen Topical System — The total of two TK-254RX per day for 5 days (one patch applied to left and right lower leg above ankle)
  Arms: TK-254RX
Drug: Flurbiprofen tablet — 3 tablets per day for 4 days
  Arms: Tablet (reference product)

SUMMARY:
This study is a single-center, open-label, multiple-dose trial performed in a 2-period, 2- sequence-cross-over design in healthy volunteers. The primary purpose of this study is to assess non-superiority of the bioavailability of TK-254RX compared with that of a marketed oral flurbiprofen-containing tablet formulation in healthy volunteers in a 2-period, 2- sequence-cross-over design and evaluate adhesion of TK-254RX. Secondary purpose is to assess safety of TK-254RX and residual amount of the patch.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 years to 64 years (inclusive)
* body-mass index (BMI): ≥18.5 kg/m² and ≤ 30.0 kg/m²
* good state of health
* non-smoker or ex-smoker for at least 3 months
* written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical triall

Exclusion Criteria:

* existing cardiac and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient
* existing or history of hypertension and/or heart failure
* existing hepatic and/or renal diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredient
* existing gastrointestinal diseases or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient
* history of gastrointestinal bleeding or perforation related to previous NSAID therapy
* active, or history of ulcerative colitis, Crohn's disease, peptic ulceration or gastrointestinal haemorrhage
* existing metabolic, endocrine and/or immunologic diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredient
* diabetes mellitus
* hyperlipidaemia (LDL > 4.16 mmol/l, HDL < 0.91 mmol/l, triglycerides > 2.28 mmol/l, cholesterol > 6.24 mmol/l)
* history of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
* presence or history of acute or chronic diseases of the skin (e.g., atopic dermatitis (eczema), neurodermatitis, contact allergy, psoriasis, vitiligo, melanoma, squamous cell carcinoma), any dermatological condition or skin sensitivity which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient
* existing or history of bronchial asthma
* known allergic reactions (e.g., bronchospasm, rhinitis, angioedema, or urticaria) to the active ingredients used, to acetylsalicylic acid or other NSAIDs, or to constituents of the pharmaceutical preparations
* history of severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the investigator
* fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase insufficiency
* galactose intolerance or Lapp lactase deficiency
* systolic blood pressure < 90 or > 139 mmHg
* diastolic blood pressure < 60 or > 89 mmHg
* heart rate < 50 bpm or > 90 bpm
* QTc interval > 450 ms for men and > 470 ms for women
* laboratory values out of normal range unless the deviation from normal is judged as not relevant for the clinical trial by the investigator
* ASAT > 20% ULN, ALAT > 10% ULN, bilirubin > 20% ULN (except in case of existing Morbus Gilbert-Meulengracht deduced from anamnesis/medical history) and creatinine > 0.1 mg/dL ULN (limit of > 0.1 mg/dL correspondents to > 9 µmol/l ULN)
* positive anti-HIV-test (if positive to be verified by western blot), HBs-AG-test or anti-HCV-test
* vaccination against COVID-19 within the last 4 weeks prior to individual intended IMP administration
* skin abnormality (e.g., tattoo (including tattoo that was removed), scar, sunburn, or obvious difference in skin colour), open sores, or excessive hair at the application sites
* acute or chronic diseases which may interfere with the pharmacokinetics of the IMP
* history of or current drug or alcohol dependence
* positive alcohol or drug test at screening examination
* regular intake of alcoholic food or beverages of ≥ 24 g pure ethanol for male or ≥ 12 g pure ethanol for female per day
* subjects who are on a diet which could affect the pharmacokinetics of the active ingredient
* regular intake of caffeine containing food or beverages of ≥ 500 mg caffeine per day
* blood donation or other blood loss of more than 400 ml within the last 2 months prior to individual enrolment of the subject
* participation in a clinical trial with administration of any investigational medicinal product during the last 2 months prior to individual enrolment of the subject
* simultaneous participation in another clinical trial with active ingredients
* regular treatment with any systemically available medication (except sexual and thyroid hormones)
* subjects, who report a frequent occurrence of migraine attacks
* positive pregnancy test at screening examination
* pregnant or lactating women
* female subjects who do not agree to apply highly effective contraceptive methods (highly effective contraceptive methods)
* subject is vulnerable such as detained or committed to an institution by a court of law or by legal authorities or close affiliation with the sponsor or the investigational site (e.g., a close relative of the investigator, dependent person (e.g., employee of or student at the investigational site), employee of the sponsor or affiliates)
* subject suspected or known not to follow instructions
* subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve over 24 hours of S-flurbiprofen for TK-254RX and tablet under steady-state conditions | Day 5 to Day 6
Peak Plasma Concentration of S-flurbiprofen for TK-254RX and tablet under steady-state conditions | Day 5 to Day 6
Characterization of patch adhesion | Day 1 to Day 6
  Measuring patch adhesion area by percentage of visually by site staff with remaining patch adhered

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve over 24 hours of S-flurbiprofen for TK-254RX on Day 1 | Day 1 to Day 2
Peak Plasma Concentration of S-flurbiprofen for TK-254RX on Day 1 | Day 1 to Day 2
Time to reach Peak Plasma Concentration of TK-254RX after the first two patches application on Day 1 | Day 1
Time before first concentration value above the lower limit of quantitation of TK-254RX after the first two patches application on Day 1 | Day 1
Trough concentration of TK-254RX | 24 hours, 48 hours, 72 hours, 96 hours, 120 hours after first TK-254RX application
  minimum concentration at the end of each dosing
Trough concentration of tablet | 24 hours, 48 hours, 72 hours, 96 hours after first tablet application
  minimum concentration at the end of each dosing
Area under the plasma concentration versus time curve of R- flurbiprofen and metabolites from the last two TK-254RX application to the time point of 24 hours under steady condition | Day 5
Peak Plasma Concentration of R-flurbiprofen and metabolites under steady condition | Day 5
Minimum plasma concentration of TK-254RX under steady condition | Day 5
Time to reach Peak Plasma Concentration of TK-254RX under steady condition | Day 5
Percentage of peak trough fluction of TK-254RX under steady condition | Day 5
Average concentration at time points on Day 5 under steady condition | Day 5
Area under the plasma concentration versus time curve from the last two TK-254RX application to last measurement time point with a concentration value above lower limit of quantitation | Day 5 to Day 8
Percentage of area under the plasma concentration versus time curve extrapolated to infinity to area under the plasma concentration versus time curve from 0 hour to infinity of the last TK-254RX application | Day 5 to Day 8
Area under the plasma concentration versus time curve from 0 hour to infinity of the last TK-254RX application | Day 5 to Day 8
Concentration at the last time point with concentration value above the lower limit of quantitation of the last TK-254RX application | Day 5 to Day 8
Last time point with concentration value above the lower limit of quantitation of the last TK-254RX application | Day 5 to Day 8
Apparent terminal elimination half-life of TK-254RX | Day 5 to Day 8
Apparent terminal elimination rate constant determined by log-linear regression of TK-254RX | Day 5 to Day 8
Area under the plasma concentration versus time curve of R-flurbiprofen and metabolites over 24 hours under steady condition | Day 4 to Day 7
Peak plasma concentration of R-flurbiprofen and metabolites of tablet under steady condition | Day 4 to Day 7
Minimum plasma concentration of tablet under steady condition | Day 4 to Day 7
Time to reach Peak Plasma Concentration of tablet under steady condition | Day 4 to Day 7
Percentage of peak trough fluction of tablet under steady condition | Day 4 to Day 7
Average concentration at time points of tablet under steady condition | Day 4 to Day 7
Area under the plasma concentration versus time curve from the first tablet administration on day 4 to last measurement time point with a concentration value above lower limit of quantitation | Day 4 to Day 7
Area under the plasma concentration versus time curve from 0 hour to infinity of tablet of administration on 4th day | Day 4 to Day 7
Percentage of area under the plasma concentration versus time curve extrapolated to infinity to area under the plasma concentration versus time curve from 0 hour to infinity of tablet of administration on 4th day | Day 4 to Day 7
Concentration at the last time point with concentration value above the lower limit of quantitation of tablet of administration on 4th day | Day 4 to Day 7
Last time point with concentration value above the lower limit of quantitation of tablet of administration on 4th day | Day 4 to Day 7
Apparent terminal elimination half-life of tablet | Day 4 to Day 7
Apparent terminal elimination rate constant determined by log-linear regression of tablet | Day 4 to Day 7
Local tolerability | within 5 min after removal of each patch as well as 12 h, 24 h, and 36 h after removal of the last 2 patches on study Day 6
  Assessing the local tolerability by using the 8-point dermal response and other effects score according to FDA recommendation
Residual amount of S-flurbiprofen | Day 5 to Day 6
  residual amount of S-flurbiprofen in used patch applied on Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Nishiyama, Study Chair — Teikoku Seiyaku Co., Ltd.
Locations (1):
- SocraTec R&D GmbH Clinical Pharmacology Unit, Mainzerhofplatz 14, Erfurt, Germany

IPD SHARING:
Plan to Share IPD: No